CLINICAL TRIAL: NCT01148914
Title: The Role of Cardiac Biomarkers in Prediction of Outcome in Atrial Fibrillation Patients Undergoing Catheter Ablation
Acronym: IMPACT
Status: Completed | Type: Observational
Sponsor: Texas Cardiac Arrhythmia Research Foundation (Other)
Responsible Party: Principal Investigator, Andrea Natale, Executive medical director, Texas Cardiac Arrhythmia Research Foundation
Other Study IDs: TCAI-IMPACT
Record Dates: First submitted 2010-06-21; First posted 2010-06-22 (Estimated); Last update posted 2012-06-01 (Estimated); Status verified 2010-06

CONDITIONS: Atrial Fibrillation
Keywords: Inflammatory biomarkers; Atrial fibrillation; Catheter ablation; To assess if pre-ablation levels of inflammatory biomarkers serve as independent predictors of procedure outcome; To evaluate the inflammatory activation following catheter ablation and examine its predictive role in procedure success; To determine if a change in the baseline level of biomarkers at 3-months follow-up has any correlation with long-term outcome; To study the association of certain biomarkers with specific types of AF (paroxysmal or persistent or long standing persistent)
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Baseline level of biomarkers
  Interventions: Other: Inflammatory biomarkers

INTERVENTIONS:
Other: Inflammatory biomarkers — tTst blood samples for cardiac biomarkers at baseline, 24-hours and 3 month post-ablation

SUMMARY:
This prospective study aims;

1. To assess if pre-ablation levels of inflammatory biomarkers serve as independent predictors of procedure outcome
2. To evaluate the inflammatory activation following catheter ablation by measuring serum-biomarker levels 24-hours after the procedure and examine the predictive role in procedure success
3. To determine if a change in the baseline level of certain inflammatory biomarkers at 3-months post-ablation period has any correlation with the long-term outcome in patients with atrial fibrillation
4. To study the association of certain biomarkers with specific types of AF (paroxysmal or persistent or long standing persistent)

DETAILED DESCRIPTION:
AF is the most common arrhythmia in clinical practice, affecting > 2.3 million people in US. It increases dramatically with age and is seen in as many as 9% of individuals by the age of 80 (1). A major cause of stroke, AF is also associated with a 2-fold increase in mortality (1).

Symptomatic AF has been demonstrated to be consistently associated with elevated inflammatory activity in the atrial tissue as evidenced by the facts that AF occurs in 40% of patients following cardiac bypass surgery and 50% of patients undergoing valvular surgery (2). Recent studies have also demonstrated that elevated CRP level can increase the risk of AF up to 31% (2). Oxidative damage experienced during AF leads to myocardial necrosis which in turn induces low-grade inflammation resulting in eventual fibrosis of the atrial myocardium. Thus, inflammation can be responsible for adverse structural and electrical remodeling of the cardiac tissue which can further perpetuate the existence, maintenance, and recurrence of this arrhythmia.

Radiofrequency catheter ablation (RFCA) has evolved as a promising curative therapy for drug-refractory AF. However, the recurrence of AF after RFCA is a common clinical problem, occurring in 25-50% of patients in the follow-up period (3) and some patients undergo multiple ablation procedures before being cured of the arrhythmia. Published retrospective studies have demonstrated that systemic inflammation generated during AF ablation is associated with fewer early arrhythmia recurrences (4). Therefore, measurement of inflammatory markers within 24 hours of RFCA could be helpful in further exploration of any association between the degree of inflammatory activation and procedure outcome.

Systemic inflammatory activation is characterized by increased circulating levels of several biomarkers for prolonged periods. Thus, examination of these biomarkers at 3-months post-procedure may provide critical insight into understanding the role of inflammation in achievement of long-term success of catheter ablation in AF patients.

Rules-Based Medicine, Inc (RBM) at 3300 Duval Road Austin, TX 78759 has developed biomarker panels that have been validated to detect early signs of inflammation. RBM will process the blood samples on a preliminary panel of ~40 biomarkers which are presumed to be possible predictors of procedural outcomes in RFCA in AF patients.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-75 years
* Patients undergoing catheter ablation of atrial fibrillation
* Able and willing to give written consent

Exclusion Criteria:

* Reversible causes of AF such as pericarditis and hyperthyroidism
* Associated chronic inflammatory diseases such as chronic gingivitis or peri-odontitis, rheumatoid Arthritis, IBD including Ulcerative Colitis and Crohn's disease, Lupus, Ankylosing Spondylitis, COPD, psoriasis, vasculitis
* Patients taking long-term steroid medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Atrial fibrillation patients undergoing catheter ablation
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
To identify serum biomarkers that correlate with procedure outcome in AF patients undergoing catheter ablation | 3-months post-procedure

SECONDARY OUTCOMES:
To identify the biomarkers which correlate with different types of AF, namely paroxysmal, persistent or long-standing persistent | 3months from the date of procedure
To identify candidate biomarkers that can predict fluid retention in the immediate post-ablation period. | 24 hours from the procedure date

CONTACTS AND LOCATIONS:
Locations (1):
- St.David's Medical Center, Austin, Texas, United States